CLINICAL TRIAL: NCT06900465
Title: Pilot Evaluation of a Psychoeducation Group for Family Caregivers of Children and Adolescents With Emotional and Behavioral Disorders (CPG-CA) in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Hao YAO, Attending Psychiatrist, Shanghai Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-73
Record Dates: First submitted 2025-03-19; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Emotional and Behavioral Disorders in Children and Adolescents
Keywords: Pilot trial; Emotional and behavioral disorder; Child and adolescent; Psychoeducation; China; Psychosocial intervention; Caregiver
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study will be a waitlist-controlled randomized pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will first receive the CPG-CA intervention.
  Interventions: Behavioral: Caregiver Psychoeducation Group for Children and Adolescents with Emotional and Behavioral Disorders (CPG-CA)
- Waitlist control group (No Intervention): The waitlist control group will receive the CPG-CA intervention after the intervention group. During the waiting period, the waitlist control group will receive care as usual.

INTERVENTIONS:
Behavioral: Caregiver Psychoeducation Group for Children and Adolescents with Emotional and Behavioral Disorders (CPG-CA) — The CPG-CA intervention is a group psychoeducational internvention for family caregivers of children and adolescents with E/BDs in China. It will consist of 10 to 15 family caregivers of children and adolescents with E/BDs, meeting once a week for 1.5 to 2 hours per session, for a total of 12 sessions over a 3-month period. The sessions will cover the following themes: (1) knowledge about child and adolescent emotional and behavioral disorders; (2) coping skills for common emotional and behavioral problems in children and adolescents; (3) problem-solving skills; (4) communication skills with children and adolescents; (5) positive parenting techniques; and (6) self-care techniques. A variety of facilitation techniques will be used in the intervention, including didactic teaching, group discussion, role-playing, and homework assignment.
  Arms: Intervention group

SUMMARY:
The goal of this waitlist-controlled randomized pilot trial is to premilinariliy learn if the CPG-CA internvention, a group psychoeducational intervention for family caregivers of children and adolescents with emotional and behavioral disorders, works to relieve caregiver burden among family caregivers of children and adolescents with emotional and behavioral disorders in China. It will also learn about the acceptability of the CPG-CA intervention. The main questions it aims to answer are:

Does the CPG-CA intervention relieve caregiver burden among family caregivers of children and adolescents with emotional and behavioral disorders in China? Is the CPG-CA intervention acceptable to family caregivers of children and adolescents with emotional and behavioral disorders in China?

Researchers will compare the CPG-CA intervention to care-as-usual to see if the CPG-CA internvention works to relieve caregiver burden among family caregivers of children and adolescents with emotional and behavioral disorders in China.

Participants will receive the CPG-CA intervention or care-as-usual for 12 weeks.

DETAILED DESCRIPTION:
In China, most children and adolescents with emotional and behavioral disorders (E/BDs) are living with families. With an extreme scarcity of child and adolescent mental health care resources in China, the primary caregiving responsibility for children and adolescents with E/BDs is laid on families. However, caregiving for children and adolescents with E/BDs could be challenging, and family caregivers of children and adolescents with E/BDs often describe their caregiving experiences as exhausting and burdensome.

To date, very few interventions in China have been designed to relieve caregiver burden among family caregivers of children and adolescents with E/BDs. Therefore, this study aims to conduct a randomized, wait-list controlled pilot trial to preliminarily evaluate the feasibility and effectiveness of the CPG-CA intervention, a group psychoeducational intervention for family caregivers of children and adolescents with E/BDs, in reducing caregiver burden among family caregivers of children and adolescents with E/BDs in China. This pilot trial will lay the groundwork for a major trial that will be conducted in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Family caregivers of children and adolescents under the age of 18 with emotional and behavioral disorders;
2. The child or adolescent must have a confirmed diagnosis of an emotional or behavioral disorder, including: emotional and behavioral disorders with onset usually occurring in childhood and adolescence, mood disorders, depressive disorders, bipolar disorder, anxiety disorders, attention-deficit/hyperactivity disorder (ADHD), conduct disorder, oppositional defiant disorder, obsessive-compulsive disorder (OCD), eating disorders, schizophrenia, and addictive disorders;
3. Providing care for a child or adolescent with an emotional or behavioral disorder for at least three months;
4. Aged 18 or older;
5. Able to provide informed consent.

Exclusion Criteria:

1. Caregivers of children and adolescents with neurodevelopmental disorders (e.g., autism, intellectual disability);
2. Paid caregivers;
3. Caregivers with severe physical illnesses or mental disorders;
4. Caregivers under the age of 18;
5. Those unable to provide informed consent;
6. Caregivers who are simultaneously participating in other support groups for family caregivers of children and adolescents with emotional and behavioral disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver burden | Baseline (T0) and 3 months (T1)
  Participants' caregiver burden will be assessed using the Zarit Burden Interview (ZBI).

SECONDARY OUTCOMES:
Caregiver burden | Baseline (T0) and 6 months (T2)
  Participants' caregiver burden will be assessed using the Zarit Burden Interview (ZBI).
Caregiver burden | Baseline (T0) and 9 months (T3)
  Participants' caregiver burden will be assessed using the Zarit Burden Interview (ZBI).
Depression | Baseline (T0) and 3 months (T1)
  Participants' depression will be assessed using the Patient Health Questionnaire (PHQ).
Depression | Baseline (T0) and 6 months (T2)
  Participants' depression will be assessed using the Patient Health Questionnaire (PHQ).
Depression | Baseline (T0) and 9 months (T3)
  Participants' depression will be assessed using the Patient Health Questionnaire (PHQ).
Anxiety | Baseline (T0) and 3 months (T1)
  Participants' anxiety will be assessed using the Generalized Anxiety Disorder Scale (GAD).
Anxiety | Baseline (T0) and 6 months (T2)
  Participants' anxiety will be assessed using the Generalized Anxiety Disorder Scale (GAD).
Anxiety | Baseline (T0) and 9 months (T3)
  Participants' anxiety will be assessed using the Generalized Anxiety Disorder Scale (GAD).
Illness perception | Baseline (T0) and 3 months (T1)
  Participants' illness perception will be assessed using the Brief Illness Perception Questionnaire (BIPQ).
Illness perception | Baseline (T0) and 6 months (T2)
  Participants' illness perception will be assessed using the Brief Illness Perception Questionnaire (BIPQ).
Illness perception | Baseline (T0) and 9 months (T3)
  Participants' illness perception will be assessed using the Brief Illness Perception Questionnaire (BIPQ).
Coping style | Baseline (T0) and 3 months (T1)
  Participants' coping style will be assessed using the Simplified Coping Style Questionnaire (SCSQ).
Coping style | Baseline (T0) and 6 months (T2)
  Participants' coping style will be assessed using the Simplified Coping Style Questionnaire (SCSQ).
Coping style | Baseline (T0) and 9 months (T3)
  Participants' coping style will be assessed using the Simplified Coping Style Questionnaire (SCSQ).
Social support | Baseline (T0) and 3 months (T1)
  Participants' social support will be assessed using the Oslo Social Support Scale (OSSS).
Social support | Baseline (T0) and 6 months (T2)
  Participants' social support will be assessed using the Oslo Social Support Scale (OSSS).
Social support | Baseline (T0) and 9 months (T3)
  Participants' social support will be assessed using the Oslo Social Support Scale (OSSS).
Positive caregiving experiences | Baseline (T0) and 3 months (T1)
  Participants' positive caregiving experiences will be assessed using the Positive Aspect of Caregiving scale (PAC).
Positive caregiving experiences | Baseline (T0) and 6 months (T2)
  Participants' positive caregiving experiences will be assessed using the Positive Aspect of Caregiving scale (PAC).
Positive caregiving experiences | Baseline (T0) and 9 months (T3)
  Participants' positive caregiving experiences will be assessed using the Positive Aspect of Caregiving scale (PAC).
Feeling of hope | Baseline (T0) and 3 months (T1)
  Participants' feeling of hope will be assessed using the Herth Hope Index (HHI).
Feeling of hope | Baseline (T0) and 6 months (T2)
  Participants' feeling of hope will be assessed using the Herth Hope Index (HHI).
Feeling of hope | Baseline (T0) and 9 months (T3)
  Participants' feeling of hope will be assessed using the Herth Hope Index (HHI).
Feeling of mastery | Baseline (T0) and 3 months (T1)
  Participants' feeling of mastery will be assessed using the Pearlin Mastery Scale (PMS).
Feeling of mastery | Baseline (T0) and 6 months (T2)
  Participants' feeling of mastery will be assessed using the Pearlin Mastery Scale (PMS).
Feeling of mastery | Baseline (T0) and 9 months (T3)
  Participants' feeling of mastery will be assessed using the Pearlin Mastery Scale (PMS).
Self-stigma | Baseline (T0) and 3 months (T1)
  Participants' self-stigma will be assessed using the stigma sub-scale of the Experiences of Caregiving Inventory (ECI).
Self-stigma | Baseline (T0) and 6 months (T2)
  Participants' self-stigma will be assessed using the stigma sub-scale of the Experiences of Caregiving Inventory (ECI).
Self-stigma | Baseline (T0) and 9 months (T2)
  Participants' self-stigma will be assessed using the stigma sub-scale of the Experiences of Caregiving Inventory (ECI).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
In order to protect participants' privacy, IPD will not be shared.